CLINICAL TRIAL: NCT01105624
Title: A Four Week Study of Azithromycin Ophthalmic Solution, 1% Versus Rewetting Drops in Subjects With History and Current Complaint of Contact Lens-Related Dry Eye (CLDE)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Mike Schiewe, Associate Director, Inspire
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 041-117; P08644
Record Dates: First submitted 2010-04-15; First posted 2010-04-16 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2011-09

CONDITIONS: Contact Lens Dry Eye
MeSH Terms: interventions — tetrahydrozoline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- azithromycin ophthalmic solution, 1% (Experimental)
  Interventions: Drug: azithromycin ophthalmic solution, 1%
- rewetting drops (Experimental)
  Interventions: Drug: Visine® for Contacts®

INTERVENTIONS:
Drug: azithromycin ophthalmic solution, 1% — 1 drop BID for the first 2 days and then 1 drop QD for the remainder of treatment period (29 ± 1 day)
  Arms: azithromycin ophthalmic solution, 1%
Drug: Visine® for Contacts® — 1-2 drops QID for the treatment period (29 ± 1 day)
  Arms: rewetting drops

SUMMARY:
The primary objective of this study is to compare the duration of subject reported comfortable contact lens daily wear time in subjects with a history and current complaint of CLDE during a 29-day treatment period of azithromycin ophthalmic solution, 1%, compared to rewetting drops

ELIGIBILITY:
Inclusion Criteria:

* Have a history of and current complaint of CLDE.
* Use properly fitted daily-wear soft contact lenses.
* Able to wear contact lenses for at least 8 hours a day.
* If female, are non-pregnant or non-lactating.

Exclusion Criteria:

* Have changed brand of contact lens or care solutions within one month prior to Visit 1.
* Use extended (overnight) wear contact lenses.
* Have a clinically significant ophthalmic abnormality.
* Have had cauterization of the punctum or have had punctal plugs (silicone or collagen) inserted or removed within the 90 days prior to the screening.
* Have any active ongoing ocular infection or ocular disease.
* Have a serious medical condition which could confound study assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-03; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Subject-reported comfortable contact lens daily wear time (hours/day) at Week 4 Endpoint | 4 weeks

SECONDARY OUTCOMES:
Subject-reported comfortable contact lens daily wear time, excluding Week 4 Endpoint | 2 weeks
Subject-reported duration of total contact lens daily wear | 4 weeks
Subject-reported rating of overall eye dryness | 4 weeks
Contact Lens-Related Dry Eye Questionnaire | 4 weeks
Tear hyperosmolarity (mOsm) | 4 weeks
Habitual low-contrast visual acuity (LCVA) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Reza Haque, MD, PhD, Study Chair — Medical Monitor
Locations (1):
- The Ohio State University, College of Optometry, Columbus, Ohio, United States

REFERENCES:
- [Derived] Nichols JJ, Bickle KM, Zink RC, Schiewe MD, Haque RM, Nichols KK. Safety and efficacy of topical azithromycin ophthalmic solution 1.0% in the treatment of contact lens-related dry eye. Eye Contact Lens. 2012 Mar;38(2):73-9. doi: 10.1097/ICL.0b013e31823ff229. PMID 22157392